CLINICAL TRIAL: NCT06408324
Title: A Retrospective Study to Evaluate the Use of Thrombopoietin Receptor Agonists (TPO-ra) in Adults With Primary Immune Thrombocytopenia (ITP) in Europe
Brief Title: Evaluation of the Use of Thrombopoietin Receptor Agonists in Adults With Primary ITP in Europe
Status: Completed | Type: Observational
Sponsor: European Research Consortium on ITP (Other)
Collaborators: Fondazione Progetto Ematologia (Other)
Responsible Party: Sponsor
Other Study IDs: VERTEX 3.0
Record Dates: First submitted 2023-12-18; First posted 2024-05-10 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Primary Immune Thrombocytopenia (ITP)
Keywords: Immune Thrombocytopenia; ITP; Thrombopoietin receptor agonists; TPO-RA; Eltrombopag; Romiplostim
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this multicenter, observational, retrospective is to evaluate the standards of use of thrombopoietin receptor agonists (TPO-RA) in adult patients with primary immune thrombocytopenia (ITP), with a particular interest on phase of ITP (defined according to time when diagnosis of ITP is established in the medical records: newly diagnosed, 0-3 months; persistent, 3-12 months, and chronic, > 12 months), tolerability, safety, posology and remissions, outside controlled clinical trials.

Secondary Objectives:

To analyze the patient characteristics that could affect the choice of thrombopoietin receptor agonist for the treatment of ITP, considering specific clinical aspects (such as previous thromboembolic disease, bleeding, platelet count, surgical procedures, etc.).

To evaluate the degree of adherence to international guidelines related to the use of thrombopoietin receptor agonists in regular clinical practice.

Data will be collected through a retrospective chart review of patients with ITP who started TPO-RA treatment between January 2014 and December 2018.

DETAILED DESCRIPTION:
Objectives:

Primary Objective:

To evaluate the standards of use of TPO-RA in regular clinical practice in Europe, with a particular interest on phase of ITP (the phase of the disease will be defined according to time when diagnosis of ITP is established in the medical records: newly diagnosed, 0-3 months; persistent, 3-12 months, and chronic, > 12 months), tolerability, safety, posology and remissions, outside controlled clinical trials.

Secondary Objectives:

To analyze the patient characteristics that could affect the choice of thrombopoietin receptor agonist for the treatment of ITP, considering specific clinical aspects (such as previous thromboembolic disease, bleeding, platelet count, surgical procedures, etc.).

To evaluate the degree of adherence to international guidelines related to the use of thrombopoietin receptor agonists in regular clinical practice.

Description of study centers:

The study will be conducted in medical departments of 18 European hospitals from 6 countries (UK, Spain, Italy, Norway, France and Switzerland), 3 sites per country.

The founding members of the European Research Consortium on ITP (ERCI) will identify and select the Sites / Investigators. The sites that will participate in this project must ensure to provide all of the patient´s care for ITP and that all the information required to complete the CRF can be obtained from the site´s medical records.

Study population:

Patients who started treatment for ITP with thrombopoietin receptor agonists (romiplostim/eltrombopag) between January 2014 and December 2018.

It is estimated that approximately 350 ITP TPO-RA treated patients will be included in the study.

Observational study course:

Screening:

Each site will screen patients reviewing medical records of patients with ITP who started treatment with thrombopoietin analogues (regardless of phase of the disease) between January 2014 and December 2016. In order to prevent screening bias, the medical records will be consecutively screened by the investigators, starting with the oldest (regarding start of ITP therapy with TPO-RA), by selecting patients who started therapy with agonists on the date nearest to January 2014.

To enroll a case in this study, the patient must have initiated a TPO-RA at the specific site that recruits such patient. If a sporadic patient with ITP has been referred from the participating site to a secondary center for specialized care, the investigator should confirm that data can be fully extracted from centralized records.

Information and consent: Screened patients invited to take part in the study will be informed by the investigator or an authorized member of the team during a hospital visit or by phone. No patient will be included in the study until having been duly informed by the investigator and having signed the informed consent.

Data collection:

Each site will collect retrospectively the data from all the patients with ITP who meet the inclusion criteria and no exclusion criteria, and agree to participate in the study by signing the informed consent.

The data will be obtained in a retrospective, non-interventionist manner to meet this study's objective, by reviewing the patient's medical records. The investigator will only collect the data available in the patients' medical records; patients will have been followed up according to regular clinical practice and received treatment according to the investigator's clinical judgement. In no case shall a patient's inclusion in the study affect regular clinical practice.

Collected data:

The collected data will include variables at the time of diagnosis (bleeding, comorbidities, biological studies), treatments received before TPO-RA, variables at time of TPO-RA initiation, and following TPO-RA therapy. Considering that patients initiated TPO-RA in 2014- 2018, data will include information before date of TPO-RA initiation (diagnosis before or in 2014- 2018), and also all the information related to TPO-RA therapy and follow-up, until the date of data collection planned in 2022-2023, independently of current or active treatment with TPO-RA agents. The data will be collected into the eCRF (electronic case report form) by the designated person at each site.

Sample size:

The objective of the study is to evaluate the use of TPO-RA in adult patients with primary ITP in Europe. The incidence of ITP in Europe ranges from 1.6 to 3.9 patients per 100,000 inhabitants. Considering a finite population, in order to identify a pattern repeated in at least 35% of patients with ±5% precision and a 95% CI, a total of 350 patients have to be enrolled. Considering a 5% loss rate (patients that withdraw their consent or those with more than 20% missing information from CRF), data from a total of at least 368 patients could finally be included.

ELIGIBILITY:
Inclusion Criteria:

* Patients over age 18 when TPO-RA was started
* Diagnosis of primary immune thrombocytopenia
* Patients who started treatment for ITP with thrombopoietin receptor agonists (romiplostim/eltrombopag) between January 2014 and December 2018.

The investigators will review the medical records of patients to include those with longer follow-up in the study, meaning those who started with the agonist on the date closest to January 2014. Patients will be included in chronological order based on date of TPO-RA initiation, and signed informed consent.

- Signed Informed consent*

* An exception will be the case of deceased patients, in which the investigator will sign and date the informed consent document, and will specify the absence of the patient's signature due to death. However, in the event that the codes of the Member State that regulate the processing of personal data of deceased persons do not enable to obtain this information, the specific regulations of each State will be followed.

Exclusion Criteria:

* Patients who had participated in studies with investigational drugs when TPO-RA was started
* Patients with a diagnosis of secondary immune thrombocytopenia when TPO-RA was started

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 350 patients will be included in the study. Each site will collect data of ITP patients who meet the screening criteria and agree to participate in the study, considering that it must include patients treated with romiplostim and eltrombopag ideally with the largest follow-up, meaning those who started agonist therapy on the date closest to January 2014.
  For the selection of patients, the investigators will detect among the patients at their center (who generally will have outpatient follow-up in consultations), those who meet the inclusion criteria defined below and who do not present any exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 275 (Actual)
Dates: Start 2022-11-24 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
Evaluation of the standards of use of TPO-RA in regular clinical practice in Europe | From the first TPO-RA treatment initiated between 1 January 2014 and 31 December 2018 up to the discontinuation of the last line of treatment with TPO-RA. The maximum follow-up period could be of 10 years.
  To evaluate the standards of use of TPO-RA in regular clinical practice in Europe, with reference to phase of ITP (defined according to time when diagnosis of ITP is established in the medical records: newly diagnosed; persistent and chronic), tolerability, safety, posology and remissions, outside controlled clinical trials.
  The primary end-point is the proportion of patients achieving a complete response (platelet count of ≥100 × 109 /L) or a response (platelet count of ≥30 × 109 /L) after TPO-RA initiation and upon switching. Responses are recorded for any TPO-RA treatment initiated between 1 January 2014 and 31 December 2018 up to the discontinuation of the last line of treatment with TPO-RA.

SECONDARY OUTCOMES:
To analyze the patient characteristics that could affect the choice of TPO-RA for the treatment of ITP and to evaluate the degree of adherence to international guidelines | From the first TPO-RA treatment initiated between 1 January 2014 and 31 December 2018 up to the discontinuation of the last line of treatment with TPO-RA. The maximum follow-up period could be of 10 years.
  Secondary efficacy end-points include the proportion of patients achieving platelet count thresholds of ≥50 × 109 /L; time to platelet response; duration of platelet response; proportion of patients achieving platelet responses upon switching, and proportion and duration of treatment-free responses (TFR). TFR is defined as a sustained platelet count ≥50 × 109 /L for 6 months following cessation of TPO-RA treatment. Complete TFR is defined as sustained platelet count ≥100 × 109 /L for 6 months following cessation of TPO-RA treatment. Safety end-points include the frequency of adverse events (AEs), including hospital admission for TPO-RA-related AEs. The AEs of special interest (AESIs), include thromboembolic events, hematological malignancies or solid tumors, hepatic abnormalities and cataracts.

CONTACTS AND LOCATIONS:
Overall Officials: Maria L. Lozano, M.D., Principal Investigator — Hematology and Medical Oncology Dept. Hospital General Universitario José María Morales Meseguer
Locations (17):
- France (3):
  - Hôpital Universitaire Henri Mondor, Créteil
  - CHU Dijon - Hôpital François Mitterrand Médecine 1 - Etudes Cliniques, Dijon
  - CHU Toulouse - Hôtel-Dieu Saint-Jacques, Toulouse
- Italy (3):
  - Careggi Hospital, Florence
  - Fondazione Policlinico A. Gemelli IRCCS, Roma
  - San Bortolo Hospital, Vicenza, Vicenza
- Norway (3):
  - Bergen Hospital, Bergen
  - Oslo Hospital, Oslo
  - Østfold Hospital, Oslo
- Spain (3):
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital General Universitario de Burgos, Burgos
  - Hospital Morales Meseguer, Murcia
- Switzerland (3):
  - Basel university hospital, Basel
  - Bern university hospital, Bern
  - Lausanne University hospital, Lausanne
- United Kingdom (2):
  - Imperial College NHS Trust, London
  - University Hospitals Plymouth NHS Trust, Plymouth

IPD SHARING:
Plan to Share IPD: No